CLINICAL TRIAL: NCT01248364
Title: An Open-label, Phase II Study to Determine Acute (After the First Dose Administration) and Chronic (After 28 Days of Treatment) Effects of the Sodium-glucose Co-transporter-2 (SGLT-2) Inhibitor Empagliflozin (BI 10773) (25 mg Once Daily) on Pre and Postprandial Glucose Homeostasis in Patients With IGT and, Type 2 Diabetes Mellitus and Healthy Subjects
Brief Title: A Study to Determine Acute (After First Dose) and Chronic (After 28 Days) Effects of Empagliflozin (BI 10773) on Pre and Postprandial Glucose Homeostasis in Patients With Impaired Glucose Tolerance and Type 2 Diabetes Mellitus and Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1245.39; 2010-018708-99 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (1):
- BI 10773 Arm (Experimental): BI 10773 high dose once daily
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — BI 10773 tablets once daily high dose

SUMMARY:
An open-label, phase II study to assess the acute and chronic effects of empagliflozin (BI 10773)on fasting and postprandial glucose homeostasis in patients with IGT and type 2 diabetes mellitus and assess the acute effects of empagliflozin in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients diagnosed with IGT according to the current ADA guidelines as a two-hour glucose levels of 140 to 199 mg/dl (7.8 mmol/l to 11.1 mmol/l) on the 75-g oral glucose tolerance test (OGTT), with an OGTT performed at the time of the screening visit (Visit 1), or

   ¿ Male and female patients diagnosed with type 2 diabetes mellitus (T2DM) prior to informed consent, on diet and exercise regimen who are drug-naïve, defined as absence of any oral antihyperglycemic therapy for 12 weeks prior starting with open-label active treatment, or
2. Male and female patients diagnosed with type 2 diabetes mellitus prior to informed consent, who are pre-treated with metformin background therapy, on a stable dose of metformin of at least 1500 mg per day, unchanged for at least 12 weeks prior starting with open-label active treatment
3. HbA1c at Visit 1 (screening)

   1. for patients diagnosed of IGT and for healthy subjects: HbA1c < 6.5%
   2. for patients diagnosed of T2DM: HbA1c =6.5% and =10.5%
4. Age = 18 at Visit 1
5. BMI = 20 and = 40 Kg/m2 at Visit 1
6. For patients with antihypertensive treatment, this must be stable (with no change in dosage) within 4 weeks prior starting with open-label active treatment
7. Signed and dated written informed consent by date of Visit 1 in accordance with GCP and local legislation

   Inclusion criteria for healthy subjects:
8. Males or females matching the below mentioned criteria and otherwise healthy according to the investigator¿s assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR) and clinical laboratory tests .
9. HbA1c at Visit 1 (screening): HbA1c < 6.5%
10. Confirmed normal glucose tolerance (NGT) by OGTT
11. Age = 45 and = 55 at Visit 1.
12. BMI = 30 and = 40 Kg/m2 (Body Mass Index) at Visit 1.
13. Signed and dated written informed consent by date of Visit 1 in accordance with GCP and local legislation.

Exclusion criteria:

1. Acute coronary syndrome (non-STEMI [ST elevation myocardial infarction], STEMI, unstable AP [angina pectoris]), stroke or Transient Ischemic Attack (TIA) within 6 months prior to informed consent.
2. Uncontrolled hyperglycaemia with a glucose level > 240 mg/dl (> 13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day).
3. Any other antidiabetic drug within 12 weeks prior to starting the open-label active treatment (Visit 4) except those defined as background via inclusion criterion 1c.
4. Indication of liver disease, defined by serum levels of either Alanine Aminotransferase (ALT [SGPT]), Aspartate Aminotransferase (AST [SGOT]), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening and/or run-in phase.
5. Impaired renal function, defined as estimated Glomerular Filtration Rate (eGFR) < 60 ml/min (moderate and severe renal impairment) as determined during screening and/or run-in phase.
6. Medical history of insufficient bladder emptying (i.e. neurogenic bladder disorders).
7. Patients with an Haemoglobin (Hb) < 11.5 g/dl (for males) and Hb < 10.5 g/dl (for females) at Visit 1.
8. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption within the last 5 years.
9. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
10. For patients on metformin background therapy, the investigator must check for potential exclusion criteria according to local metformin label.
11. Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
12. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM. However, the use of inhaled steroids (e.g., for asthma, Chronic Obstructive Pulmonary Disease [COPD]) is not an exclusion as these do not cause systemic steroid action.
13. Alcohol or drug abuse (according to investigators judgment) within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake.
14. Intake of an investigational drug in another trial Participation in another trial within 30 days prior to intake of study medication in this trial.
15. Pre-menopausal women (last menstruation < = 1 year prior to informed consent) who:

    Are nursing or pregnant or Are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.
16. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- 1245.39.43001 Boehringer Ingelheim Investigational Site, Graz, Austria
- 1245.39.49002 Boehringer Ingelheim Investigational Site, Neuss, Germany
- 1245.39.39001 Boehringer Ingelheim Investigational Site, Pisa, Italy

REFERENCES:
- [Derived] Ferrannini E, Baldi S, Frascerra S, Astiarraga B, Barsotti E, Clerico A, Muscelli E. Renal Handling of Ketones in Response to Sodium-Glucose Cotransporter 2 Inhibition in Patients With Type 2 Diabetes. Diabetes Care. 2017 Jun;40(6):771-776. doi: 10.2337/dc16-2724. Epub 2017 Mar 21. PMID 28325783
- [Derived] Muscelli E, Astiarraga B, Barsotti E, Mari A, Schliess F, Nosek L, Heise T, Broedl UC, Woerle HJ, Ferrannini E. Metabolic consequences of acute and chronic empagliflozin administration in treatment-naive and metformin pretreated patients with type 2 diabetes. Diabetologia. 2016 Apr;59(4):700-8. doi: 10.1007/s00125-015-3845-8. Epub 2015 Dec 24. PMID 26704626
- [Derived] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454

RESULTS

PARTICIPANT FLOW:
Groups:
- T2DM Naive: Patients diagnosed with type 2 diabetes mellitus (T2DM) who have not been treated with any antihyperglycemic therapy for the last 12 weeks prior to the study. Patients received empagliflozin (empa) 25mg tablet once daily for 28 days.
- T2DM Metformin: Patients diagnosed with type 2 diabetes mellitus (T2DM) who are on stable dose of metformin of at least 1500 mg per day, for the last 12 weeks prior to the study. Patients received empagliflozin (empa) 25mg tablet once daily for 28 days.
- Impaired Glucose Tolerance: Patients diagnosed with impaired glucose tolerance (IGT) according to American Diabetes Association (ADA) guidelines. Patients received empagliflozin (empa) 25mg tablet once daily for 28 days.
- Healthy Subjects: Healthy subjects received a single dose of empagliflozin (empa) 25mg, in tablet form.
Period: Overall Study
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Started | 32 | 34 | 13 | 12
Completed Acute Phase:Single Dose, Day 1 | 32 | 34 | 13 | 12
Completed Chronic Phase:28-day Treatment | 32 | 33 | 13 | 0
Completed | 32 | 33 | 13 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients/healthy subjects treated with at least one dose of empagliflozin.
Groups:
- Total: Total of all reporting groups
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects | Total
Number analyzed (Participants) | 32 | 34 | 13 | 12 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.0) | 63.3 (6.5) | 50.8 (9.8) | 47.7 (2.3) | 58.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 5 | 2 | 28
  Male | 21 | 24 | 8 | 10 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Plasma Glucose at Day 1
Description: Change from baseline of Fasting Plasma glucose (FPG) 3 hours and 35 minutes before meal at day 1
Time Frame: Baseline and day 1
Population: Treated set which included all patients/healthy subjects with at least one dose of empagliflozin (original result (OR))
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 34 | 13 | 12
mmol/L | 0.20 (0.12) | 0.39 (0.13) | -0.96 (0.86) | -0.47 (0.97)
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.2790, ANCOVA; Based on ANCOVA with terms for baseline FPG, diagnosis group, and baseline FPG by diagnosis group interaction; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.16 to 0.55], Standard Error of Mean 0.18 — Difference calculated as T2DM metformin minus T2DM Naive

2. Primary Outcome: Change From Baseline in Fasting Plasma Glucose at Day 28
Description: Change from baseline of Fasting Plasma glucose (FPG) 3 hours and 35 minutes before meal at day 28.
  Note, healthy subjects only received a single dose of empa so assessments at day 28 are not applicable
Time Frame: Baseline and day 28
Population: Treated set, which included all patients/healthy subjects with at least one dose of empagliflozin (original result (OR)), for patients who completed the day 28 visit
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 33 | 13 | 0
mmol/L | -1.02 (0.13) | -0.79 (0.15) | -0.81 (1.12) |
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.2438, ANCOVA; Based on ANCOVA with terms for baseline FPG, diagnosis group and baseline FPG by diagnosis group interaction; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.16 to 0.62], Standard Error of Mean 0.20 — Difference calculated as T2DM metformin minus T2DM Naive

3. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: Fast, at Day 1
Description: Change from baseline in rate of endogenous glucose production (EGP) fast after one dose
Time Frame: Baseline and day 1
Population: Treated set (OR)
Measure: Least Squares Mean (Standard Error); unit: umol/kgFFM/min
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 34 | 13 | 12
umol/kgFFM/min | 4.21 (0.45) | 4.51 (0.60) | 3.28 (0.89) | 1.10 (0.97)
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.6931, ANCOVA; Based on ANCOVA with terms for baseline EPG fast, diagnosis group and baseline EPG fast by diagnosis group interaction; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-1.19 to 1.79], Standard Error of Mean 0.75 — Difference calculated as T2DM metformin minus T2DM Naive

4. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: Fast, at Day 28
Description: Change from baseline in rate of endogenous glucose production (EGP) fast after 28 days of treatment.
  Note, healthy subjects only received a single dose of empa so assessments at day 28 are not applicable.
Time Frame: Baseline and day 28
Population: Treated set (OR) for patients who completed the day 28 visit
Measure: Least Squares Mean (Standard Error); unit: umol/kgFFM/min
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 33 | 13 | 0
umol/kgFFM/min | 2.79 (0.71) | 4.63 (0.86) | 1.47 (1.44) |
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.1028, ANCOVA; Based on ANCOVA with terms for baseline EPG fast, diagnosis group and baseline EPG fast by diagnosis group interaction; Mean Difference (Final Values) = 1.84, 95% CI 2-sided [-0.38 to 4.07], Standard Error of Mean 1.12 — Difference calculated as T2DM metformin minus T2DM Naive

5. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: AUC 5h, at Day 1
Description: Change from baseline in the area under the curve of endogenous glucose production (EGP) from 0 to 5 hours (EGP AUC 5h) after meal.
Time Frame: 0 minutes (min), 15min, 30min, 45min, 1hour (h), 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 4h 30min and 5h after meal at baseline and day 1
Population: Treated set (OR)
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 34 | 13 | 11
g | 3.28 (1.80) | 8.76 (1.77) | 3.70 (2.73) | 9.22 (3.94)
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.0326, ANCOVA; Based on ANCOVA with terms for baseline EPG AUC 5h, diagnosis group and baseline EPG AUC 5h by diagnosis group interaction; Mean Difference (Final Values) = 5.48, 95% CI 2-sided [0.47 to 10.50], Standard Error of Mean 2.52 — Difference calculated as T2DM metformin minus T2DM Naive

6. Primary Outcome: Change From Baseline in Glucose Metabolism (Pre-meal and Postprandial Glucose), PPG iAUC 5h, at Day 1
Description: Change from baseline in the incremental area under the curve of postprandial plasma glucose from 0 to 5 hours (PPG iAUC 5h), defined as the area under the curve of timepoints 0 to 5 hours after meal reduced by the pre-meal plasma glucose at 0 hours.
Time Frame: as for outcome 5
Population: Treated set (OR)
Measure: Least Squares Mean (Standard Error); unit: g/dL/h
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 34 | 13 | 11
g/dL/h | -1.94 (0.53) | -3.52 (0.61) | -5.49 (1.95) | -9.20 (3.91)
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.0552, ANCOVA; Based on ANCOVA with terms for baseline PPG iAUC 5h, diagnosis group and baseline PPG iAUC 5h by diagnosis group interaction; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-3.20 to 0.04], Standard Error of Mean 0.81 — Difference calculated as T2DM metformin minus T2DM Naive

7. Primary Outcome: Change From Baseline in Glucose Metabolism (Pre-meal and Postprandial Glucose), PPG iAUC 5h, at Day 28
Description: Change from baseline in the incremental area under the curve of postprandial plasma glucose from 0 to 5 hours (PPG iAUC 5h), defined as the area under the curve of timepoints 0 to 5 hours after meal reduced by the pre-meal plasma glucose at 0 hours.
  Note, healthy subjects only received a single dose of empa so assessments at day 28 are not applicable.
Time Frame: 0 minutes (min), 15min, 30min, 45min, 1hour (h), 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 4h 30min and 5h after meal at baseline and day 28
Population: Treated set (OR) for patients who completed the day 28 visit
Measure: Least Squares Mean (Standard Error); unit: g/dL/h
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 33 | 13 | 0
g/dL/h | -0.71 (0.67) | -0.40 (0.72) | -7.31 (2.91) |
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.7561, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-1.66 to 2.27], Standard Error of Mean 0.99 — Difference calculated as T2DM metformin minus T2DM Naive

8. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: AUC 5h, at Day 28
Description: Change from baseline in the area under the curve of endogenous glucose production (EGP) from 0 to 5 hours (EGP AUC 5h) after meal.
  Note, healthy subjects only received a single dose of empa so assessments at day 28 are not applicable.
Time Frame: as for outcome 7
Population: Treated set (OR) for patients who completed the day 28 visit
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 33 | 13 | 0
g | 1.89 (1.35) | 5.02 (1.33) | 3.14 (2.35) |
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.1024, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 3.13, 95% CI 2-sided [-0.64 to 6.90], Standard Error of Mean 1.89 — Difference calculated as T2DM metformin minus T2DM Naive

9. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: iAUC 5h, at Day 1
Description: Change from baseline in the incremental area under the curve of endogenous glucose production from 0 to 5 hours (EGP iAUC 5h), defined as the area under the curve of timepoints 0 to 5 hours after meal reduced by the pre-meal endogenous glucose production at 0 hour.
Time Frame: 0 minutes (min), 15min, 30min, 45min, 1hour (h), 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 4h 30min and 5h after drug administration at baseline and day 1
Population: Treated set (OR)
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 34 | 13 | 11
g | -8.52 (1.79) | -7.22 (2.33) | -3.75 (3.82) | 1.28 (4.80)
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.6576, ANCOVA; Based on ANCOVA with terms for baseline EPG iAUC 5h, diagnosis group and baseline EPG iAUC 5h by diagnosis group interaction; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-4.53 to 7.14], Standard Error of Mean 2.93 — Difference calculated as T2DM metformin minus T2DM Naive

10. Secondary Outcome: Change From Baseline in Rate of Endogenous Glucose Production: iAUC 5h, at Day 28
Description: Change from baseline in the incremental area under the curve of endogenous glucose production from 0 to 5 hours (EGP iAUC 5h), defined as the area under the curve of timepoints 0 to 5 hours after meal reduced by the pre-meal endogenous glucose production at 0 hour.
  Note, healthy subjects only received a single dose of empa so assessments at day 28 are not applicable.
Time Frame: 0 minutes (min), 15min, 30min, 45min, 1hour (h), 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 4h 30min and 5h after drug administration at baseline and day 28
Population: Treated set (OR) for patients who completed the day 28 visit
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Number analyzed (Participants) | 32 | 33 | 13 | 0
g | -6.95 (2.26) | -10.63 (2.50) | -0.49 (5.22) |
Statistical Analysis 1: Comparison: T2DM Naive vs T2DM Metformin; No formal testing, exploratory analysis only; Test type: Superiority or Other; p = 0.2795, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-10.41 to 3.05], Standard Error of Mean 3.38 — Difference calculated as T2DM metformin minus T2DM Naive

ADVERSE EVENTS:
Time Frame: From first intake of study drug until 7 days after the last treatment intake, 5 weeks
Groups:
- Healthy Subjects: Healthy subjects received empagliflozin (empa) 25mg tablet once daily for 28 days.
Arm/Group | T2DM Naive | T2DM Metformin | Impaired Glucose Tolerance | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/34 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/32 | 5/34 | 4/13 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T2DM Naive (N=32) | T2DM Metformin (N=34) | Impaired Glucose Tolerance (N=13) | Healthy Subjects (N=12)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T2DM Naive (N=32) | T2DM Metformin (N=34) | Impaired Glucose Tolerance (N=13) | Healthy Subjects (N=12)
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.